CLINICAL TRIAL: NCT05254054
Title: The Effect of Whole Body Vibration on Dynamic Knee Stability in Patients After Anterior Cruciate Ligament Reconstruction
Brief Title: The Effect of Whole Body Vibration After ACLR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Xin He, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019.432
Record Dates: First submitted 2022-01-27; First posted 2022-02-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: ACL Injury
Keywords: ACL; dynamic knee stability; whole body vibration
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: This is a randomized control trial. Participants will be randomly allocated into either intervention group(vibration training+ conventional rehabilitation program) or control group(conventional rehabilitation program).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration group (Experimental): Participants in Vibration group will receive an 8-week whole body vibration training in addition to conventional exercise training.
  Interventions: Other: whole body vibration; Other: Conventional exercise training
- Control group (Active Comparator): Participants in Vibration group will only receive conventional exercise training.
  Interventions: Other: Conventional exercise training

INTERVENTIONS:
Other: whole body vibration — The whole body vibration is used when vibrations (mechanical oscillations) of a certain frequency are transferred to the human body. Humans are exposed to vibration through a contact surface that is in a mechanical vibrating state. It has been considered as an alternative and safe method for neuromuscular training and may be incorporated into current neuromuscular rehabilitation programs so as to enhance muscle recovery
  Arms: Vibration group
Other: Conventional exercise training — A set of conventional exercises designed for ACL rehabilitation

SUMMARY:
This is a randomised clinical trial to detect the effect of an 8-week whole body vibration training on muscle function and dynamic knee function during single leg squat and single leg hop in patients after anterior cruciate ligament reconstruction

DETAILED DESCRIPTION:
In Hong Kong, over 3000 cases of ACL reconstruction are operated annually to restore knee stability. Despite recovery of knee passive laxity and muscle strength, dynamic knee stability is often not restored. The whole body vibration has been found to improve muscle strength, proprioception and balance after ACL reconstruction. This project will investigate the effect of whole body vibration on muscle elasticity, muscle coordination and landing knee biomechanics. It may provide useful evidence to the application of whole body vibration in improving dynamic knee stability, which will lead to a significant improvement in healthcare management for ACL patients . The current study serves to provide a clinical guideline for post-ACL reconstruction rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-50;
2. Physically active before injury with Tegner score more than 6 (recreational/professional sport level);
3. Scheduled for ACLR because of sport injury;
4. Be able to walk with a pair of elbow crutches independently at 1 month after ACLR.

Exclusion Criteria:

1. Concomitant posterior cruciate ligament or lateral collateral ligament injury in the same knee;
2. Injury to the contralateral side;
3. Medical problems that are contradictory to WBV;
4. Prior experience of WBV to avoid any training or memory effect;
5. Women with pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
knee flexion angle | immediately after intervention, three month after intervention
  Peak value of knee flexion will be assessed by the skin marker-based motion analysis system (Vicon MX, Oxford, UK) during single leg squat and single leg hop landing.
knee valgus angle | immediately after intervention, three month after intervention
  Peak value of knee valgus will be assessed by the skin marker-based motion analysis system (Vicon MX, Oxford, UK) during single leg squat and single leg hop landing.
knee internal rotation angle | immediately after intervention, three month after intervention
  Peak value of knee internal rotation will be assessed by the skin marker-based motion analysis system (Vicon MX, Oxford, UK) during single leg squat and single leg hop landing.
Vertical ground reaction force | immediately after intervention, three month after intervention
  Peak vertical ground reaction force will be evaluated by a synchronized force plate during single leg hop landing.
Knee valgus torque | immediately after intervention, three month after intervention
  Peak knee valgus torque will be evaluated by a synchronized force plate during single leg hop landing.
Knee extension torque | immediately after intervention, three month after intervention
  Peak knee extension torque will be evaluated by a synchronized force plate during single leg hop landing.

SECONDARY OUTCOMES:
muscle strength | immediately after intervention, three month after intervention
  Isometric muscle strength of quadriceps and hamstring will be tested using an hand-held dynamometer. The isokinetic muscle strength of quadriceps and hamstring will be tested at 60°/s and 180°/s by the isokinetic dynamometer
muscle elasticity | immediately after intervention, three month after intervention
  Shear elastic modulus of vastus medialis, vastus lateralis, semimembranosus and biceps femoris will be assessed by shear wave elastography ultrasound.
muscle activation | immediately after intervention, three month after intervention
  Muscle activity level of vastus lateralis, vastus medialis, biceps femoris and semitendinosus will be assessed by electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Xin He, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No